CLINICAL TRIAL: NCT00449566
Title: Magnetic Resonance Imaging of Brain Development in Autism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Other Study IDs: METC 05/208-K
Record Dates: First submitted 2007-03-18; First posted 2007-03-20 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Autism
Keywords: Magnetic Resonance Imaging; Diffusion Tensor Imaging
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate brain development in autism by longitudinally assessing children with autism, as well as typically developing controls, using advanced MR techniques. We will use longitudinal diffusion tensor imaging (DTI) measures to investigate the protracted development of long-range white matter fibers in autism. In addition, we will investigate the effect of autism risk genes on brain development.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 - 18 years at initial MRI

Inclusion criteria for subjects with autism

1) DSM-IV (APA, 1994) diagnosis of autism, according to ADI-R interview

Inclusion criteria for controls

1. no DSM-IV (APA, 1994) diagnosis, according to DISC interview
2. no scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)
3. IQ > 70

Exclusion Criteria:

1. major illness of the cardiovascular, the endocrine, the pulmonal or the gastrointestinal system
2. presence of metal objects in or around the body (pacemaker, dental braces)
3. history of or present neurological disorder
4. for individuals over 12 years of age: legal incompetence, defined as the obvious inability to comprehend the information that is presented by the investigator and is outlined in the Information letter and on which the decision to participate in the study is to be based

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Durston, Ph.D., Principal Investigator — Rudolf Magnus Institute of Neuroscience, University Medical Center Utrecht; Herman van Engeland, M.D. Ph.D., Study Chair — Rudolf Magnust Institute of Neuroscience, UMC Utrecht
Locations (1):
- Dept. of Child and Adolescent Psychiatry, UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Langen M, Durston S, Staal WG, Palmen SJ, van Engeland H. Caudate nucleus is enlarged in high-functioning medication-naive subjects with autism. Biol Psychiatry. 2007 Aug 1;62(3):262-6. doi: 10.1016/j.biopsych.2006.09.040. Epub 2007 Jan 16. PMID 17224135
- See also: Lab homepage with info for subjects (in Dutch) — http://www.niche-lab.nl